CLINICAL TRIAL: NCT02655627
Title: Can Internet Based Exercise Training Be an Alternative to Supervised Group Exercise Training in Patients With Type 2 Diabetes?
Brief Title: Internet Based Exercise Training in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Collaborators: Istanbul University (Other)
Responsible Party: Principal Investigator, Buket AKINCI, PT, MSc, Biruni University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014/1977
Record Dates: First submitted 2016-01-12; First posted 2016-01-14 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 DM; internet based exercise training; group exercise training; glycemic control
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (3):
- Group A (Experimental): Usual Care Group: A brochure which emphasis the importance of physical activity and exercise in Type 2 DM will be given to the patients in this group after the evaluation.
  Interventions: Other: Physical activity counselling via a brochure
- Group B (Experimental): Supervised Clinical Exercise Training Group: Patients in this group will continue group exercise training includes aerobic and resistance training, 1 hour in a day, 3 times in a week for 8 weeks with the supervision of a researcher physiotherapist.
  Interventions: Other: group exercise training
- Group C (Experimental): Internet Based Exercise Training Group. the patients to this group will be a member of the web site named www.diyabetvehareket.com. The participation of the patients will be provided with the videos directing them to 1 hour in a day, 3 times in a week for 8 week both aerobic and resistance exercise training from the researcher physiotherapist.
  Interventions: Other: Internet based exercise training

INTERVENTIONS:
Other: Internet based exercise training
  Arms: Group C
Other: group exercise training
  Arms: Group B
Other: Physical activity counselling via a brochure
  Arms: Group A

SUMMARY:
Type 2 Diabetes Mellitus (DM) is a disease which is characterized with insulin resistance and exercise has positive effects on glycemic control and cardiovascular disease (CVD) development in these patients. Encouraging physical activity and exercise with using internet-based technology provides; potential to reach more people via comparatively low cost, 24 hour accessibility to services and for clinician, more frequent communication ability with the patient. In literature, there is no study examined exercise training via internet in patients with Type 2 DM. For this reason, considering the lack of the literature, the investigators aimed to compare the effects of internet based combined exercise training on glycemic control, functional capacity and physical activity level with supervised group training in patients with Type 2 DM. The purpose of the study is to provide convenience of rehabilitation access, glycemic control, offer an alternative physiotherapy and rehabilitation service which can help to improve physical activity level and obtain quantitative data for the applicability and contribution of internet based exercise training in patients with Type 2 DM.

ELIGIBILITY:
Inclusion Criteria:

* HbA1c level between %6,5-11
* Patients who can reach 420 meters in 6 minutes walking test
* Patients who are available high speed internet from home, work or mobile phone

Exclusion Criteria:

* Non-Cooperation

  * Uncontrolled Hypertension and cardiac arrythmia
  * Severe neurological and pulmonary disorder
  * Patients who had Percutan Transluminal Coronary Angiography or cardiac pacemaker
  * Previous Myocardial Infarction
  * Previous amputation
  * Major musculoskeletal problem
  * Chronic renal failure
  * Patients who had hip or knee prothesis within 5 years
  * Diabetic ulceration pr neuropathy
  * Pregnancy
  * Breastfeeding
  * Hemolytic anemia
* Renal anemia

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-09-01 (Actual)

PRIMARY OUTCOMES:
HbA1c | 2 months

SECONDARY OUTCOMES:
fasting blood glucose | 2 months
Body fat ratio | 2 months
Body Muscle Ratio | 2 months
6 minute walking distance | 2 months
International Physical Activity Questionnaire | 2 months
Number of Steps (Mean of 7 days) | 2 months
Quadriceps Muscle Strength (for left and right) | 2 months
Euro Quality of Life-5 Dimension | 2 months

OTHER OUTCOMES:
cholesterol levels | 2 months

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Buket AKINCI, Istanbul
  - Istanbul University, Istanbul